CLINICAL TRIAL: NCT02926573
Title: Perioperative Gabapentin Use In Head And Neck Mucosal Surgery Patients: A Randomized Clinical Trial
Brief Title: Perioperative Gabapentin Use In Head And Neck Mucosal Surgery Patients
Acronym: GABA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201605121
Record Dates: First submitted 2016-09-26; First posted 2016-10-06 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer; Acute Pain; Postoperative Pain
Keywords: oral cavity; oropharynx; hypopharynx and larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Acute Pain; Pain, Postoperative; Laryngeal Diseases | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Active Comparator): Gabapentin liquid by mouth or Per Tube 300mg twice a day
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo liquid by mouth or Per Tube twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin
  Arms: Gabapentin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Patient satisfaction with healthcare is increasingly being utilized as a metric to reflect provider and hospital quality of care. Furthermore, at the core of a healthcare team and healthcare system is the desire to provide patients with the best possible care in order to achieve the best possible outcomes. Providers have the duty to identify areas of needed improvement within the domains of treatment. An area of need that is ubiquitous within medicine is pain control; in this case acute postoperative pain control is the targeted condition. Studies have already shown that better control of acute postoperative pain leads to shortened hospital stays, reduced hospital costs and patient morbidity, improved patient satisfaction and a reduced likelihood of developing chronic pain. Research within the field of pain management has definitively revealed that a combination of different medication regimens can control acute postoperative pain better than narcotics alone. In particular, the medication gabapentin has been shown to improve acute postop pain in many kinds of surgical settings, and it is a safe medication with arguably fewer side effects than narcotics. The investigators know that certain groups of post surgical otolaryngology patients can be at risk for high levels of postoperative pain. Given all of this information, physicians have a responsibility to utilize medications such as gabapentin to do a better job of controlling patient's pain. This investigation is a quality improvement project designed to elucidate the benefits of gabapentin in pain management in patients undergoing surgery of the head and neck mucosal surfaces. It will provide much needed data in an understudied population and ultimately will improve the practice of pain management, patient satisfaction and quality of care delivered in the Barnes otolaryngology department.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing definitive mucosal head and neck resection including oral cavity, oropharynx, larynx, and hypopharynx
* At least one night of planned inpatient stay

Exclusion Criteria:

* Incapable of giving informed consent
* Age less than 18
* Glomerular Filtration Rate (GFR) less than 30
* Allergy to gabapentin
* Baseline gabapentin or lyrica use
* Chronic opioid use for over six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Townsend, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Townsend M, Liou T, Kallogjeri D, Schoer M, Scott-Wittenborn N, Lindburg M, Bottros M, Jackson RS, Nussenbaum B, Piccirillo JF. Effect of Perioperative Gabapentin Use on Postsurgical Pain in Patients Undergoing Head and Neck Mucosal Surgery: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2018 Nov 1;144(11):959-966. doi: 10.1001/jamaoto.2018.0282. PMID 29710075
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 06/24/2016 and closed to participant enrollment on 06/30/2017.
Pre-assignment Details: 13 participants were enrolled but withdrew prior to study participation with no medication given. 8 participants withdrew due to patient preference and 5 withdrew due to cancellation of surgery.
Period: Overall Study
Arm/Group | Gabapentin | Placebo
Started | 55 | 55
Completed | 44 | 46
Not Completed | 11 | 9
Not completed — Nausea | 1 | 0
Not completed — Remain intubated | 2 | 2
Not completed — Change in surgery plan | 3 | 1
Not completed — Change to outpatient status | 5 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Return to operating room | 0 | 2
Not completed — Delirium | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11.3) | 60.9 (10.0) | 61.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 33 | 36 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 44 | 46 | 90
Participant's opinion on effectiveness of narcotic pain medication [Count of Participants; unit: Participants] — Population: Some participants were not included as they had never had narcotic pain medication prior to surgery.
  Participants
    Low effectiveness: number analyzed (Participants) | 37 | 42 | 79
    Low effectiveness | 8 | 10 | 18
    High effectiveness: number analyzed (Participants) | 37 | 42 | 79
    High effectiveness | 29 | 32 | 61
Participant's experience with significant amount of daily pain [Count of Participants; unit: Participants] — Participants were asked about daily pain aside from the pain due to the current head and neck condition. Population: 3 responses are missing because surveys were not given (1 in the gabapentin arm and 2 in the placebo arm)
  Participants
    number analyzed (Participants) | 43 | 44 | 87
    No daily pain | 40 | 36 | 76
    Daily pain | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Daily Narcotic Consumption
Description: Total amount of narcotic use in morphine equivalents will be divided by the total hours of inpatient hospitalization, multiplied by 24 hours, to obtain the daily narcotic consumption.
Time Frame: Daily from date of randomization until post-op day 2 or date of discharge, whichever comes first.
Measure: Median (Full Range); unit: mg/hour
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 44 | 46
mg/hour | 1.60 [0 to 6.11] | 1.59 [0 to 5.84]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; Median Difference (Final Values) = 0.26, 95% CI 2-sided [-0.27 to 0.94]

2. Secondary Outcome: Patient Reported Post-treatment Pain Satisfaction as Measured by How Often the Participant's Pain Was Well Controlled
Description: -A discharge survey to document patient satisfaction and perceived pain control was given at the time of the last VAS score.
Time Frame: Once on post-op day 2 or day of discharge, whichever comes first
Population: The participants who did not answer this question on the survey were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 43
Participants
  Never | 1 | 0
  Sometimes | 1 | 6
  Usually/Always | 40 | 37
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; Percent Difference = 9.2, 95% CI 2-sided [-3.0 to 21]

3. Secondary Outcome: Patient Reported Post-treatment Pain Satisfaction as Measured by How Often the Hospital Staff Did Everything They Could do to Help the Participant's Pain
Description: as for outcome 2
Time Frame: Once on post-op day 2 or day of discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 43
Participants
  Never | 0 | 0
  Sometimes | 0 | 2
  Usually | 5 | 5
  Always | 37 | 36

4. Secondary Outcome: Patient Reported Post-treatment Pain Satisfaction as Measured by Overall Pain Control
Description: as for outcome 2
Time Frame: Once on post-op day 2 or day of discharge, whichever comes first
Measure: Count of Participants; unit: Participants
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 43
Participants
  Very satisfied | 30 | 34
  Somewhat satisfied | 7 | 5
  Neutral | 2 | 0
  Somewhat dissatisfied | 0 | 2
  Dissatisfied | 3 | 2
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; Percent Difference = -2, 95% CI 2-sided [-15 to 11] — The estimation parameter is based on those participants who answered they were "very satisfied" with overall pain control

5. Secondary Outcome: Mean Pain With Resting Score as Measured by VAS
Description: * Subjective pain scores were captured using the Visual Analog Scale (VAS). Subjects were asked to "Please rate your current pain level with no movement (rest), with a cough, and with a swallow". Subjects marked a point on a 100-mm line anchored "no pain" on the left end and "worst possible pain" on the right end.
  * Pain literature reports that scores in the 10-30mm range correlate clinically with mild pain, in the 30-60 or 70mm range with moderate pain, and in the >70 range with severe pain
Time Frame: Baseline through post operative day 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 43
mm
  Post-operative Day 1 7AM | 44 (26.9) | 46 (24.9)
  Post-operative Day 1 10AM | 29 (26.5) | 37 (28.2)
  Post-operative Day 1 7PM | 25 (25.3) | 32 (25.9)
  Post-operative Day 2 7AM | 27 (26.2) | 32 (24.5)
  Post-operative Day 2 10AM | 23 (23.3) | 30 (22.4)
  Post-operative Day 2 7PM | 25 (24.3) | 33 (25.7)
  Post-operative Day 3 7AM | 22 (22.4) | 32 (26.1)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [-3.4 to 18.3] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 7AM
Statistical Analysis 2: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [-2.9 to 20.3] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 10AM
Statistical Analysis 3: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 7.2, 95% CI 2-sided [-4.6 to 18.9] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 7PM
Statistical Analysis 4: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [-6.6 to 16.8] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 7AM
Statistical Analysis 5: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [-3.6 to 18.3] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 10AM
Statistical Analysis 6: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 8.0, 95% CI 2-sided [-5.6 to 21.6] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 7PM
Statistical Analysis 7: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 10.1, 95% CI 2-sided [-3.5 to 23.8] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 3 7AM

6. Secondary Outcome: Mean Pain With Coughing Score as Measured by VAS
Description: as for outcome 5
Time Frame: Baseline through post operative day 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 43
mm
  Post-operative Day 1 7AM | 36 (27.9) | 46 (26.7)
  Post-operative Day 1 10AM | 36 (30.0) | 45 (28.2)
  Post-operative Day 1 7PM | 34 (26.5) | 41 (27.4)
  Post-operative Day 2 7AM | 34 (27.0) | 39 (27.6)
  Post-operative Day 2 10AM | 28 (23.3) | 39 (28.5)
  Post-operative Day 2 7PM | 30 (25.1) | 45 (29.7)
  Post-operative Day 3 7AM | 27 (24.1) | 39 (27.1)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 10.7, 95% CI 2-sided [-0.9 to 22.3] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 7AM
Statistical Analysis 2: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 9.1, 95% CI 2-sided [-3.4 to 21.6] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 10AM
Statistical Analysis 3: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [-6.1 to 18.6] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 7PM
Statistical Analysis 4: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-7.3 to 17.8] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 7AM
Statistical Analysis 5: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 11.2, 95% CI 2-sided [-1.4 to 23.8] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 10AM
Statistical Analysis 6: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 14.9, 95% CI 2-sided [-0.1 to 29.9] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 7PM
Statistical Analysis 7: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 11.6, 95% CI 2-sided [-2.8 to 26.0] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 3 7AM

7. Secondary Outcome: Mean Pain With Swallowing Score as Measured by VAS
Description: as for outcome 5
Time Frame: Baseline through post operative day 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Gabapentin | Placebo
Number analyzed (Participants) | 42 | 43
mm
  Post-operative Day 1 7AM | 49 (32.3) | 48 (30.7)
  Post-operative Day 1 10AM | 46 (33.8) | 51 (31.3)
  Post-operative Day 1 7PM | 41 (29.2) | 52 (28.5)
  Post-operative Day 2 7AM | 41 (30.1) | 48 (28.9)
  Post-operative Day 2 10AM | 37 (29.5) | 45 (29.8)
  Post-operative Day 2 7PM | 40 (29.3) | 56 (29.3)
  Post-operative Day 3 7AM | 35 (28.0) | 52 (30.5)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-14.7 to 11.9] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 7AM
Statistical Analysis 2: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-8.6 to 19.2] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 10AM
Statistical Analysis 3: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 10.9, 95% CI 2-sided [-2.4 to 24.2] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 1 7PM
Statistical Analysis 4: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 7.0, 95% CI 2-sided [-6.6 to 20.7]; This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 7AM
Statistical Analysis 5: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 8.0, 95% CI 2-sided [-6.4 to 22.3] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 10AM
Statistical Analysis 6: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 15.7, 95% CI 2-sided [-0.4 to 31.7] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 2 7PM
Statistical Analysis 7: Comparison: Gabapentin vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 16.7, 95% CI 2-sided [0.0 to 33.4] — This statistical analysis is for the mean difference between the 2 arms at Post-Operative Day 3 7AM

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the day of surgery to the end of the study which is post-operative day 3 or sooner if discharge is sooner than post-operative day 3.
Arm/Group | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 1/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 46/55 | 50/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gabapentin (N=55) | Placebo (N=55)
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute renal failure (Renal and urinary disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 2
Airway bleed (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Airway edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 3
Allergic contact dermatitis (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 32 | 35
Anxiety (Psychiatric disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrioventricular block (Cardiac disorders) | 1 | 0
Bleeding at wound site (Injury, poisoning and procedural complications) | 0 | 1
Bloody sputum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blurry vision (Eye disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 6 | 7
Chest pain (Cardiac disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Congestive heart failure exacerbation (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Delerium (Psychiatric disorders) | 2 | 0
Delirium/alcohol withdrawal (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3
Diplopia (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 6 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Elevated alkaline phosphatase (Investigations) | 0 | 1
Elevated liver enzymes (Investigations) | 1 | 0
Elevated white blood cells (Blood and lymphatic system disorders) | 29 | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Eye tingling (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fever (General disorders) | 1 | 3
Flap necrosis (Injury, poisoning and procedural complications) | 1 | 1
Hematochezia (Gastrointestinal disorders) | 1 | 0
Hematoma (Vascular disorders) | 3 | 2
Hematoma at flap site (Injury, poisoning and procedural complications) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Hemorrhage at resection site (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 11 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 3
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 37 | 40
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 14 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 9 | 9
Hypoparathyroidism (Endocrine disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 14 | 6
Hypotension (Vascular disorders) | 7 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Iatrogenic bradycardia (Cardiac disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Laryngeal hemorrhage (Gastrointestinal disorders) | 0 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Left arm surgical site cellulitis (Infections and infestations) | 1 | 0
Left neck numbness (Nervous system disorders) | 1 | 0
Left shoulder weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Left upper extremity swelling (General disorders) | 1 | 0
Microcytic anemia (Blood and lymphatic system disorders) | 1 | 0
Myasthenia gravis exacerbation (Nervous system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3
Neck fistula (General disorders) | 0 | 1
Neck hematoma (Vascular disorders) | 1 | 1
Neck infection (Infections and infestations) | 0 | 1
Nonsustained ventricular tachycardia (Cardiac disorders) | 0 | 1
Oral wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Oropharyngeal bleeding (Gastrointestinal disorders) | 1 | 0
Orthostasis (Vascular disorders) | 1 | 0
Oxygen desaturation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Parasthesia (right foot) (Nervous system disorders) | 1 | 0
Pharyngeal leak (Gastrointestinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pressure ulcer - coccyx (Skin and subcutaneous tissue disorders) | 1 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rectal bleeding (Gastrointestinal disorders) | 0 | 1
Reflux (Gastrointestinal disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Right upper extremity tingling (Nervous system disorders) | 0 | 1
Sensation of reflux/burning with tube feeds (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 14 | 12
Stoma bleeding (General disorders) | 1 | 0
Stoma dehiscence (Gastrointestinal disorders) | 1 | 0
Superficial dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Superior thryroid artery bleed hematemesis (Injury, poisoning and procedural complications) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Surgical site infection (MRSA) (Infections and infestations) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 1
Thrombosis (Vascular disorders) | 2 | 0
Tongue edema (Gastrointestinal disorders) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 | 3
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 3
Weight loss (Investigations) | 0 | 1
Wound breakdown (Injury, poisoning and procedural complications) | 1 | 1
Wound infection (Infections and infestations) | 1 | 2
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Hypochloremia (Metabolism and nutrition disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
All subjects were analyzed following intention to treat principles and were included in the final analysis if greater than one night of admission was achieved before study participation ended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT02926573/Prot_SAP_000.pdf